CLINICAL TRIAL: NCT03728777
Title: Resveratrol Supplementation in Patients With Mitochondrial Myopathies and Skeletal Muscle Fatty Acid Oxidation Disorders: A Double-blind, Placebo-controlled, Cross Over Study
Brief Title: Resveratrol Supplementation in Patients With Mitochondrial Myopathies and Skeletal Muscle Fatty Acid Oxidation Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Nicoline Løkken, Medical Doctor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H-17039503
Record Dates: First submitted 2018-04-19; First posted 2018-11-02 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Mitochondrial Myopathies; Fatty Acid Oxidation Defects
MeSH Terms: conditions — Mitochondrial Myopathies | interventions — Resveratrol

STUDY DESIGN:
Intervention Model Description: double-blind, randomized, placebo-controlled, cross-over study.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Resveratrol
- Resveratrol (Experimental): Over the counter supplement
  Interventions: Dietary Supplement: Resveratrol

INTERVENTIONS:
Dietary Supplement: Resveratrol — Resveratrol supplementation 1000 mg /day or placebo

SUMMARY:
The purpose of this study is to investigate the potential beneficial effects of a daily supplement of Resveratrol (1000mg/day) on physical ability and on muscle metabolism in patients with verified mitochondrial myopathy and patients with a verified fatty acid oxidation defect of VLCAD and CPTII deficiencies. Investigators hypothesize an improved muscle metabolism, mitochondrial function, fatty acid oxidation and thus improvement of physical ability.

DETAILED DESCRIPTION:
Study design: double-blind, randomized, placebo-controlled, cross-over study.

To ensure enough participants, and due to the risk of a heterogeneous cohort, a cross-over design is chosen, where participants are their own controls. 10 patients with mitochondrial myopathy and 10 patients with fatty acid oxidation defects will be included. Eligible patients will be randomized using a 1:1 assignment ratio to receive placebo or RSV first. Each treatment will be administered orally twice daily for 8 weeks, followed by a 4 weeks wash-out, and afterwards a new 8-week treatment period.

During the 20-week trial period, subjects will visit the trial site on five occasions, for functional assessments (cycle ergometer testing), blood sampling and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is willing and able to provide written informed consent prior to participation.
2. Patient is ≥18 and ≤80 years of age at baseline.
3. Patients have genetically verified mitochondrial disorder or a fatty acid oxidation deficiency (VLCAD/CPTII).
4. Patient has a clinical presentation, signs or symptoms suggestive of myopathy (e.g., easy fatigability, exercise intolerance, muscle pain) in the opinion of the Investigator.
5. Patient is ambulatory.

Exclusion Criteria:

1. Patient has any prior or current medical conditions that, in the judgment of the Investigator, would prevent the patient from safely participating in and/or completing all study requirements.
2. Patient has symptoms of mitochondrial myopathy due to known secondary mitochondrial dysfunction (e.g., drug-induced myopathy).
3. Patient does not have the cognitive capacity to understand/comprehend and complete all study assessments.
4. Pregnancy or breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Heart rate | 20 weeks
  Decrease in heart rate during constant load cycling exercise.

SECONDARY OUTCOMES:
Peak oxygen utilization | 20 weeks
  VO^2max (ml/min)
Fatty acid oxidation | 20 weeks
  Fatty acid oxidation will be assessed by stable isotope technique (only for fatty acid oxidation defect disease subgroup)
Perceived exertion | 20 weeks
  Evaluation of perceived exertion (Borg score) during constant workload cycling
Fatigue Severity Scale score | 20 weeks
  Evaluation of self-rated fatigue
SF-36 questionnaire | 20 weeks
  Evaluation of self-rated daily function scores

CONTACTS AND LOCATIONS:
Overall Officials: John Vissing, professor, Study Director — Copenhangen Neuromuscular Center, Rigshospitalet, Denmark
Locations (1):
- Copenhagen Neuromuscular Center, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided